CLINICAL TRIAL: NCT01364818
Title: Characterization of Potential Biomarkers to Assess Brain Connectivity in Neurodevelopmental Disorders in Response to Treatment
Brief Title: Brain Connectivity in Neurodevelopmental Disorders in Response to Treatment
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Linmarie Sikich, MD, Associate Professor, University of North Carolina, Chapel Hill
Other Study IDs: 11-0962
Record Dates: First submitted 2011-05-16; First posted 2011-06-02 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Autism Spectrum Disorders; Psychosis; Fragile X Syndrome
MeSH Terms: conditions — Autism Spectrum Disorder; Psychotic Disorders; Fragile X Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Placebo Comparator: Placebo: No treatment/ performance of somatosensory task (cortical metrics) without any intervention. The somatosory task will be performed before any intervention/at the midpoint/ and finally at the end.
- Active Comparator: Active Medication: Treatment (memantine, lurasidone)/ performance of somatosensory task (cortical metrics) with intervention. The somatosory task will be performed before any intervention has started/at the midpoint/ and finally at the end.

SUMMARY:
The purpose of the proposed research is to study the potential changes in biomarkers of patients with neurodevelopmental disorders in response to treatment in clinical trials or in private psychiatry practice utilizing non-invasive psychophysiological measurements. The investigators plan to obtain psychophysical measurements throughout several periods of treatment.

DETAILED DESCRIPTION:
This study will employ a non-invasive custom-built four-point vertical displacement stimulator. This is used to deliver sinusoidal vibrations at very low amplitudes (0-400 microns) to the tips of the fingers. The forearm of the subject rests on the stimulator, the finger tips are vibrated, and the subject answers questions prompted by a computer monitor about their perception of the stimuli. Research staff may explain questions and prompts in a way that may be better understood by the subjects if the subjects experience any difficulty.

This device will be used to obtain objective psychophysical measurements as subjects undergo treatment. The investigators hope that this study will eventually assist in the long term goal of studying ways to develop diagnostic methods, based on changes in cortical information processing capabilities that occur with neurodevelopmental disorders. This would enable clinicians to more objectively determine prognosis and the best course of intervention for their patients.

This study will consent up to 60 subjects who are have initiated or changed pharmacologic treatment as either a participant in a clinical trial or as a private patient of one of the study doctors. Subjects who are a participant in another clinical trial may be one an active medication or a non-active medication(placebo). Subjects will have 7 visits in this study (w0 prior to initiating new treatment, and 4,8, 26 52,78 and 104 weeks after starting the the new treatment. The latter visits may occur either while the individual is taking the medication or after the individual has stopped treatment (in order to assess persistence of treatment-related changes).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are eligible to participate in a clinical trial conducted by Dr. Sikich or individuals who have initiated/changed pharmacologic treatment (as private patient of a study physician)
* Diagnosis of autism spectrum disorder (ASD), psychotic spectrum disorder (PSD), or Fragile X syndrome.
* Ages 3-45 inclusive

Exclusion Criteria:

• Non-English Speaking subject or parent/guardian

Ages: 3 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants recruited for a clinical trial conducted by Dr. Sikich, or are private patients of one of the study doctors.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pre-Post Treatment Differences between Groups | Subjects' V1 occurs within 2 wks of start of tx, V2 within 2 wks of tx midpt, V3 within 1 wk of end of tx. V4 will occur at Mo. 6, V5 will occur at Mo. 12, V6 will occur at Mo. 18, V7 will occur at Mo. 24/End of Study.
  The primary analyses will examine whether the pre-post treatment difference in the effect of confounding stimuli (eg. ratio of confounded stimuli/control stimuli) on amplitude discrimination varies between the two groups (active treatment, no active treatment group) using an unpaired t test.

CONTACTS AND LOCATIONS:
Overall Officials: Linmarie Sikich, M.D., Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No